CLINICAL TRIAL: NCT03088345
Title: Use of Arginine Vasopressin in Early Postoperative Management After Fontan Palliation
Brief Title: Early Use of Vasopressin in Post-Fontan Management
Acronym: VAMP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Amee Bigelow, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRBNet 885148
Record Dates: First submitted 2017-02-28; First posted 2017-03-23 (Actual); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Circulatory Perfusion Disorder; Congenital Heart Disease; Single-ventricle
Keywords: Fontan Palliation Surgery; Post-Operative Care
MeSH Terms: conditions — Heart Defects, Congenital; Univentricular Heart | interventions — Arginine Vasopressin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vasopressin, Arginine (Experimental): Patients randomized to this arm will receive a continuous arginine vasopressin in normal saline carrier infusion immediately following the modified ultrafiltration (MUF) period of their cardiac surgery.
  Interventions: Drug: Vasopressin, Arginine
- Placebo (Placebo Comparator): Patients randomized to this arm will receive a continuous normal saline carrier infusion immediately following the modified ultrafiltration (MUF) period of their cardiac surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vasopressin, Arginine — Subjects will be started on a blinded continuous infusion of study drug/placebo in the OR, immediately following the completion of the MUF at 0.3 mU/kg/min. All caregivers will be blinded to the arm assignment. The infusion will run for 20 hours, at which time it will be weaned off at 0.1 mU/hr, over 3 hours.During the active study period, the care team will treat subjects per SOC, using any preferred medication to correct low cardiac output; there is no restriction on using open-label vasopressin during the active study treatment period.
  Other Names: Arginine Vasopressin
  Arms: Vasopressin, Arginine
Drug: Placebo — Subjects will be started on a blinded continuous infusion of study drug/placebo in the OR, immediately following the completion of the MUF at 0.3 mU/kg/min. All caregivers will be blinded to the arm assignment. The infusion will run for 20 hours, at which time it will be weaned off at 0.1 mU/hr, over 3 hours.During the active study period, the care team will treat subjects per SOC, using any preferred medication to correct low cardiac output; there is no restriction on using open-label vasopressin during the active study treatment period.
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
This is an investigator initiated, prospective, single-center, double-blinded, randomized, placebo-controlled trial of post-operative low dose vasopressin infusions as an early treatment of low systemic perfusion in pediatric patients following Fontan palliation.

DETAILED DESCRIPTION:
The treatments for preventing and managing low cardiac output syndrome after congenital heart surgery with cardiopulmonary bypass include manipulations of vascular volume and infusions of phosphodiesterase inhibitors (milrinone) and catecholamines (epinephrine and norepinephrine) for inotropic and vasoactive effects, all of which have associated risks which can contribute to morbidity and mortality. Vasopressin, a vasoactive drug with efficacy in septic shock, has also been utilized to improve postoperative hemodynamics after cardiac surgery in children. It is a common institutional practice to use vasopressin in this patient population, but usually after escalation through two or three other vasoactive drugs. There have been several studies in pediatrics and adults which suggest that vasopressin is not inferior to other vasoconstrictor therapies, and advantageous when looking at specific end points. The investigators propose to randomize the use of vasopressin to use at an earlier point in our typical post-operative medication strategy. The proposed study is a double blinded, randomized, placebo control study of vasopressin infusion immediately after the completion Fontan operation. The goal is to identify a vasoactive treatment strategy that improves hemodynamics with lower catecholamine infusion burden, reduces volume of fluid resuscitation, and reduces in-hospital resource utilization.

Neonatal and pediatric interventions associated with congenital heart disease (CHD) continue to produce improved outcomes. There are no established guidelines for managing patients after congenital heart surgery due to lesion-specific unique challenges in the post-operative period. Volume resuscitation and catecholamine infusions are the traditional treatment methods to maintain adequate perfusion. However, these two treatment modalities are associated with increased risk of worsening lung function and prolonged ventilator support with aggressive fluid resuscitation, increased myocardial oxygen demand, and precipitation of arrhythmias. Given the multifactorial etiology of postoperative low cardiac output syndrome, it is often unclear which catecholamine infusion is optimal to improve circulatory function. Vasopressin, an alternative vasoactive therapy commonly utilized in shock, has been utilized to improve postoperative hemodynamics in neonatal and pediatric patient populations and has recently gained more attention.

The use of arginine vasopressin infusion in infants and children after cardiac surgery was first reported in 1999 in a case series of 11 patients with vasodilatory shock in the postoperative period. This case series reported initiation of vasopressin for hypotension refractory to traditional treatment methods and reported a significant rise in hemodynamics with improved blood pressure in all patients as well as weaning inotropic support in 10/11 patients. Since this study there have been conflicting reports regarding vasopressin levels and the use of vasopressin to improve hemodynamics. Results from a study published in 2008 evaluated vasopressin levels in 39 patients with CHD in the pre and post-operative periods and concluded that children do not have deficient levels of vasopressin following surgery with cardiopulmonary bypass (CPB). In addition, lower levels were not associated with hypotension. A larger study in 2010 of 121 patients who had congenital heart surgery with CPB described results suggestive of clinically important hypotension associated with low vasopressin levels. Several other publications have reported improved blood pressure and decreased catecholamine usage in patients with CHD. Two of these reports have focused on vasopressin use in infants with single ventricle physiology. In all of these reported case series the vasopressin infusion has been initiated in the post-operative period as a rescue therapy. None of the studies have advocated for initiation of vasopressin immediately post-operatively and prior to a time period of hemodynamic instability, except for one retrospective chart review by Alten et al. This study from 2012 initiated vasopressin in the operating room after CPB in 19 neonates undergoing either an arterial switch for d-transposition of the great arteries or the Norwood palliation procedure for hypoplastic left heart syndrome. In this study, all neonates in whom vasopressin was initiated in the operating room received significantly lower amounts of volume replacement and catecholamine support in the immediate post-operative period. They also described lower heart rate, lower incidence of arrhythmias, shorter duration of mechanical ventilation and shorter intensive care unit stay when compared to lesion-matched control group. More recently in 2016, a single center retrospectively reviewed their experience with vasopressin and patients undergoing Fontan operations over a 10 year period and it's effects on chest tube output. They determined that patients receiving vasopressin perioperatively had less chest tube output and shorter duration of chest tube drainage in addition to shorter hospital length of stay and improved fluid balance as compared to historical controls.

There is a gap in the literature describing improved outcomes with a specific targeted vasoactive and inotropic therapy regimen to use in the post-operative Fontan procedure patients. This proposed novel study will further provide evidence for outcome based post-operative medical interventions. The proposed study is a double blinded, randomized control study of vasopressin infusion versus placebo in the first 24-hours after Fontan completion. The aim of this study is to evaluate the impact of vasopressin on the early postoperative course in a relatively homogenous population, with specific attention to catecholamine use, hemodynamics, pleural drainage, extracardiac organ function (kidney and liver) and length of stay. Furthermore, the investigators plan to evaluate vasopressin levels between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Planned completion of Fontan palliation
* English or Spanish speaking
* Completion of Informed Consent

Exclusion Criteria:

* Previous failed attempts at Fontan completion with subsequent takedown
* Planned concomitant atrioventricular valvuloplasty or neoaortic valve or arch reconstruction at the time of Fontan completion
* History of renal failure requiring renal replacement therapy
* Absence of informed consent

Ages: 3 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Hoffman, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Delmas A, Leone M, Rousseau S, Albanese J, Martin C. Clinical review: Vasopressin and terlipressin in septic shock patients. Crit Care. 2005 Apr;9(2):212-22. doi: 10.1186/cc2945. Epub 2004 Sep 9. PMID 15774080
- [Background] Leibovitch L, Efrati O, Vardi A, Matok I, Barzilay Z, Paret G. Intractable hypotension in septic shock: successful treatment with vasopressin in an infant. Isr Med Assoc J. 2003 Aug;5(8):596-8. No abstract available. PMID 12929303
- [Background] Tsuneyoshi I, Yamada H, Kakihana Y, Nakamura M, Nakano Y, Boyle WA 3rd. Hemodynamic and metabolic effects of low-dose vasopressin infusions in vasodilatory septic shock. Crit Care Med. 2001 Mar;29(3):487-93. doi: 10.1097/00003246-200103000-00004. PMID 11373409
- [Background] Rosenzweig EB, Starc TJ, Chen JM, Cullinane S, Timchak DM, Gersony WM, Landry DW, Galantowicz ME. Intravenous arginine-vasopressin in children with vasodilatory shock after cardiac surgery. Circulation. 1999 Nov 9;100(19 Suppl):II182-6. doi: 10.1161/01.cir.100.suppl_2.ii-182. PMID 10567301
- [Background] Hall LG, Oyen LJ, Taner CB, Cullinane DC, Baird TK, Cha SS, Sawyer MD. Fixed-dose vasopressin compared with titrated dopamine and norepinephrine as initial vasopressor therapy for septic shock. Pharmacotherapy. 2004 Aug;24(8):1002-12. doi: 10.1592/phco.24.11.1002.36139. PMID 15338849
- [Background] Gaies MG, Gurney JG, Yen AH, Napoli ML, Gajarski RJ, Ohye RG, Charpie JR, Hirsch JC. Vasoactive-inotropic score as a predictor of morbidity and mortality in infants after cardiopulmonary bypass. Pediatr Crit Care Med. 2010 Mar;11(2):234-8. doi: 10.1097/PCC.0b013e3181b806fc. PMID 19794327
- [Background] Gaies MG, Jeffries HE, Niebler RA, Pasquali SK, Donohue JE, Yu S, Gall C, Rice TB, Thiagarajan RR. Vasoactive-inotropic score is associated with outcome after infant cardiac surgery: an analysis from the Pediatric Cardiac Critical Care Consortium and Virtual PICU System Registries. Pediatr Crit Care Med. 2014 Jul;15(6):529-37. doi: 10.1097/PCC.0000000000000153. PMID 24777300
- [Background] Argenziano M, Choudhri AF, Oz MC, Rose EA, Smith CR, Landry DW. A prospective randomized trial of arginine vasopressin in the treatment of vasodilatory shock after left ventricular assist device placement. Circulation. 1997 Nov 4;96(9 Suppl):II-286-90. PMID 9386112
- [Background] Landry DW, Levin HR, Gallant EM, Ashton RC Jr, Seo S, D'Alessandro D, Oz MC, Oliver JA. Vasopressin deficiency contributes to the vasodilation of septic shock. Circulation. 1997 Mar 4;95(5):1122-5. doi: 10.1161/01.cir.95.5.1122. PMID 9054839
- [Background] Landry DW, Levin HR, Gallant EM, Seo S, D'Alessandro D, Oz MC, Oliver JA. Vasopressin pressor hypersensitivity in vasodilatory septic shock. Crit Care Med. 1997 Aug;25(8):1279-82. doi: 10.1097/00003246-199708000-00012. No abstract available. PMID 9267938
- [Background] Kampmeier TG, Rehberg S, Westphal M, Lange M. Vasopressin in sepsis and septic shock. Minerva Anestesiol. 2010 Oct;76(10):844-50. PMID 20935620
- [Background] Dunser MW, Mayr AJ, Ulmer H, Ritsch N, Knotzer H, Pajk W, Luckner G, Mutz NJ, Hasibeder WR. The effects of vasopressin on systemic hemodynamics in catecholamine-resistant septic and postcardiotomy shock: a retrospective analysis. Anesth Analg. 2001 Jul;93(1):7-13. doi: 10.1097/00000539-200107000-00003. PMID 11429329
- [Background] Jerath N, Frndova H, McCrindle BW, Gurofsky R, Humpl T. Clinical impact of vasopressin infusion on hemodynamics, liver and renal function in pediatric patients. Intensive Care Med. 2008 Jul;34(7):1274-80. doi: 10.1007/s00134-008-1055-2. Epub 2008 Mar 19. PMID 18350274
- [Background] Tweddell JS, Nersesian M, Mussatto KA, Nugent M, Simpson P, Mitchell ME, Ghanayem NS, Pelech AN, Marla R, Hoffman GM. Fontan palliation in the modern era: factors impacting mortality and morbidity. Ann Thorac Surg. 2009 Oct;88(4):1291-9. doi: 10.1016/j.athoracsur.2009.05.076. PMID 19766824
- [Background] Hirsch JC, Goldberg C, Bove EL, Salehian S, Lee T, Ohye RG, Devaney EJ. Fontan operation in the current era: a 15-year single institution experience. Ann Surg. 2008 Sep;248(3):402-10. doi: 10.1097/SLA.0b013e3181858286. PMID 18791360
- [Background] Meyer DB, Zamora G, Wernovsky G, Ittenbach RF, Gallagher PR, Tabbutt S, Gruber PJ, Nicolson SC, Gaynor JW, Spray TL. Outcomes of the Fontan procedure using cardiopulmonary bypass with aortic cross-clamping. Ann Thorac Surg. 2006 Nov;82(5):1611-8; discussion 1618-20. doi: 10.1016/j.athoracsur.2006.05.106. PMID 17062214
- [Background] Evora PR, Pearson PJ, Schaff HV. Arginine vasopressin induces endothelium-dependent vasodilatation of the pulmonary artery. V1-receptor-mediated production of nitric oxide. Chest. 1993 Apr;103(4):1241-5. doi: 10.1378/chest.103.4.1241. PMID 8131474
- [Background] Sai Y, Okamura T, Amakata Y, Toda N. Comparison of responses of canine pulmonary artery and vein to angiotensin II, bradykinin and vasopressin. Eur J Pharmacol. 1995 Aug 25;282(1-3):235-41. doi: 10.1016/0014-2999(95)00343-j. PMID 7498282
- [Background] Novella S, Martinez AC, Pagan RM, Hernandez M, Garcia-Sacristan A, Gonzalez-Pinto A, Gonzalez-Santos JM, Benedito S. Plasma levels and vascular effects of vasopressin in patients undergoing coronary artery bypass grafting. Eur J Cardiothorac Surg. 2007 Jul;32(1):69-76. doi: 10.1016/j.ejcts.2007.03.047. Epub 2007 May 15. PMID 17507236
- [Background] Morrison WE, Simone S, Conway D, Tumulty J, Johnson C, Cardarelli M. Levels of vasopressin in children undergoing cardiopulmonary bypass. Cardiol Young. 2008 Apr;18(2):135-40. doi: 10.1017/S1047951108001881. Epub 2008 Mar 7. PMID 18325140
- [Background] Mastropietro CW, Rossi NF, Clark JA, Chen H, Walters H 3rd, Delius R, Lieh-Lai M, Sarnaik AP. Relative deficiency of arginine vasopressin in children after cardiopulmonary bypass. Crit Care Med. 2010 Oct;38(10):2052-8. doi: 10.1097/CCM.0b013e3181eed91d. PMID 20683257
- [Background] Lechner E, Hofer A, Mair R, Moosbauer W, Sames-Dolzer E, Tulzer G. Arginine-vasopressin in neonates with vasodilatory shock after cardiopulmonary bypass. Eur J Pediatr. 2007 Dec;166(12):1221-7. doi: 10.1007/s00431-006-0400-0. Epub 2007 Jan 16. PMID 17225160
- [Background] Mastropietro CW, Clark JA, Delius RE, Walters HL 3rd, Sarnaik AP. Arginine vasopressin to manage hypoxemic infants after stage I palliation of single ventricle lesions. Pediatr Crit Care Med. 2008 Sep;9(5):506-10. doi: 10.1097/PCC.0b013e3181849ce0. PMID 18679141
- [Background] Alten JA, Borasino S, Toms R, Law MA, Moellinger A, Dabal RJ. Early initiation of arginine vasopressin infusion in neonates after complex cardiac surgery. Pediatr Crit Care Med. 2012 May;13(3):300-4. doi: 10.1097/PCC.0b013e31822f1753. PMID 21926664

RESULTS

PARTICIPANT FLOW:
Groups:
- Vasopressin, Arginine: Patients randomized to this arm will receive a continuous arginine vasopressin infusion immediately following the modified ultrafiltration (MUF) period of their cardiac surgery.
  Vasopressin, Arginine: Subjects will be started on a blinded continuous infusion of study drug/placebo in the OR, immediately following the completion of the MUF at 0.3 mU/kg/min. All caregivers will be blinded to the arm assignment. The infusion will run for 20 hours, at which time it will be weaned off at 0.1 mU/hr, over 3 hours.During the active study period, the care team will treat subjects per SOC, using any preferred medication to correct low cardiac output; there is no restriction on using open-label vasopressin during the active study treatment period.
- Placebo: Patients randomized to this arm will receive a continuous normal saline infusion immediately following the modified ultrafiltration (MUF) period of their cardiac surgery.
  Placebos: Subjects will be started on a blinded continuous infusion of study drug/placebo in the OR, immediately following the completion of the MUF at 0.3 mU/kg/min. All caregivers will be blinded to the arm assignment. The infusion will run for 20 hours, at which time it will be weaned off at 0.1 mU/hr, over 3 hours.During the active study period, the care team will treat subjects per SOC, using any preferred medication to correct low cardiac output; there is no restriction on using open-label vasopressin during the active study treatment period.
Period: Overall Study
Arm/Group | Vasopressin, Arginine | Placebo
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vasopressin, Arginine | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: months] | 40 (23) | 37 (7) | 38 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 7 | 8 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Hemodynamics as Characterized by Vasoactive Inotrope Score (VIS)
Description: The vasoactive inotrope score (VIS) is a linear sum of vasoactive and inotrope durg infusion doses. It is usually reported as dimensionless but is sometimes reported as normalized to dopamine mcg/kg/min equivalents. The score starts at 0 and has no defined upper limit, with a commonly observed range 0-50. It is used as a measure of the intensity of hemodynamic support, with higher scores indicating more vasoactive drug support for patients. The relationship of VIS to other patient outcomes is not consistent. It will be calculated hourly for all subjects and compared between groups over the entire observation timeframe.
Time Frame: 48 hours post-operative
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Vasopressin, Arginine | Placebo
Number analyzed (Participants) | 10 | 10
units | 11 (1.6) | 11.3 (1.9)

2. Primary Outcome: Hemodynamics as Characterized by Mean Arterial Pressure
Description: Organ perfusion pressure measured as Mean Arterial Pressure (MAP). It will be measured hourly for 24 postoperative hours for all subjects and compared between the two study groups over the whole time of observation as the main between-group effect in panel regression.
Time Frame: 24 hours post-operative
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Vasopressin, Arginine | Placebo
Number analyzed (Participants) | 10 | 10
mmHg | 67 (1.3) | 66 (1.1)

3. Primary Outcome: Hemodynamics as Characterized by Transpulmonary Pressure Gradient
Description: The transpulmonary pressure gradient (TPG), defined as the difference between mean pulmonary arterial pressure (Ppa) and left/common atrial (common atrial) pressure (Pla) will be measured hourly for 24 postoperative hours for all subjects and compared between the two study groups over the whole time of observation as the main between-group effect in panel regression.
Time Frame: 24 hours post-operative
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Vasopressin, Arginine | Placebo
Number analyzed (Participants) | 10 | 10
mmHg | 6.4 (0.5) | 8.3 (0.5)

4. Secondary Outcome: Renal Dysfunction as Characterized by Change in Cystatin Level
Description: Cystatin levels will be measured at baseline (immediately before cardiopulmonary bypass) 24 hours postoperative. The change (postoperative minus baseline) in cystatin level will be compared between groups.
Time Frame: from baseline pre-cardiopulmonary bypass to 24 hours post-operative
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Vasopressin, Arginine | Placebo
Number analyzed (Participants) | 10 | 10
mg/L | 0.095 [-0.086 to 0.277] | 0.017 [-0.160 to 0.194]

5. Secondary Outcome: Liver Dysfunction as Characterized by Transaminase Levels
Description: Transaminase levels (alanine and aspartate, measured in IU/L ) will be tracked for all patients and changes will be compared between study groups.
Time Frame: 48 hours post-operative
Measure: Mean (Standard Deviation); unit: iU/L
Arm/Group | Vasopressin, Arginine | Placebo
Number analyzed (Participants) | 10 | 10
iU/L | 715 (653) | 522 (397)

6. Other Pre Specified Outcome: Resource Utilization Measured by Length of Stay (LOS)
Description: Length of stay (LOS) measured in postoperative hours compared between groups
Time Frame: from time of operation until hospital discharge
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Vasopressin, Arginine | Placebo
Number analyzed (Participants) | 10 | 10
hours | 180 (72) | 203 (72)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Vasopressin, Arginine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
The study design represents experience at a single center and may have limited generalizability. This study was underpowered to detect differences in many clinical outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT03088345/Prot_SAP_000.pdf